CLINICAL TRIAL: NCT01883830
Title: "Feasibility and Efficacy of Virtual Reality With Xbox Kinect in the Rehabilitation of Cronic Traumatic Brain Injuries: a Randomized Controlled Trial".
Brief Title: Xbox in the Rehabilitation of Chronic Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, Physical Medicine and Rehabilitation doctor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kinect_study; Kinect (Other: Ferrara University Hospital)
Record Dates: First submitted 2013-04-05; First posted 2013-06-21 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Traumatic Brain Injury; Balance Disorders; Attention Deficits
Keywords: traumatic brain injury (TBI); balance disorders; attention deficits; x-box; gaming; virtual reality
MeSH Terms: conditions — Brain Injuries, Traumatic; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gaming therapy (Xbox) (Experimental): Subjects belonging to the first group will receive a gaming therapy protocol using the Xbox console. They will receive 24 sessions of treatment within 8 weeks (3 sessions per week). Patients will be required to concentrate in games whose major purposes are increasing balance, selective attention and attention shifting. During sessions the patient will be carefully controlled by a researcher who will prevent the risk of falling and impulsiveness reactions.
  Interventions: Device: gaming therapy (Xbox)
- Dynamic balance platform training (Active Comparator): Control group will receive the same amount of therapy (24 sessions) using a dynamic balance platform (Biodex).
  Interventions: Device: Dynamic balance platform (Biodex)

INTERVENTIONS:
Device: gaming therapy (Xbox)
  Arms: gaming therapy (Xbox)
Device: Dynamic balance platform (Biodex)
  Arms: Dynamic balance platform training

SUMMARY:
Traumatic brain injury is an extremely common disease, it counts 50.000 deaths and 235.000 hospitalizations every year. Functional consequences of an acquired brain injury have a considerable impact on quality of lives of patients and care-givers with direct effects on balance, mobility and on psycho-social functions. Attention deficits are one of the most frequent and disabling consequences of severe brain injury. Within the wide spectrum of attentive problems, patients with traumatic brain injury frequently have shown difficulties in divided attention. Patients, care-givers and professionals frequently refer difficulties also in selective attention and vigilance as consequence of the trauma. It has been shown how these difficulties are tightly related with the missed return to work after two years from the injury.

The hypothesis of this study is to investigate the feasibility of a rehabilitative protocol on gaming using the console Xbox and its efficacy in improving balance, mobility, risk of falling, attentive functions (selective and divided attention) in subjects which have had a traumatic brain injury at least 12 months before.

DETAILED DESCRIPTION:
Inclusion Criteria:

Chronic traumatic brain injury (>12 months) Age>18, <70 years old Presence of a moderate balance deficit identified by CB&M with a score < 65 or presence of a selective attention and shifting attention deficit identified by the TEA computerized battery (Tau<37).

ELIGIBILITY:
Inclusion Criteria:

* Chronic traumatic brain injury (>12 months)
* Age>18, <70 years old
* Presence of a moderate balance deficit identified by UBS with a score>15 and < 60 or presence of a selective attention and shifting attention deficit identified by the TEA computerized battery (Tau<37).

Exclusion Criteria:

* Neurologic diseases associated with possible involvement of motor functions
* Medical conditions that could interfere with the safe conclusion of the study protocol
* Severe cognitive-behavioural diseases (LCF<6),
* severe psychiatric diseases
* Use of walking aids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in balance with Community Balance & Mobility Scale (CB&M) | 1)A week prior to treatment beginning 2) the week after treatment 3)three months follow up.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) | 1)A week prior to treatment beginning 2) the week after treatment 3)three months follow up.
Unified Balance Scale (UBS) | 1)A week prior to treatment beginning 2) the week after treatment 3)three months follow up.
Participation Objective, Participation Subjective Scale(POPS) | 1)A week prior to treatment beginning 2) the week after treatment 3)three months follow up.
postural sway | 1)A week prior to treatment beginning 2) the week after treatment 3)three months follow up.
  Center of pressure (COP) trajectories
Attentive functions evaluation Attentive functions evaluation | 1)A week prior to treatment beginning 2) the week after treatment 3)three months follow up.
  TEA computerized battery

CONTACTS AND LOCATIONS:
Overall Officials: Nino Basaglia, MD, Principal Investigator — Ferrara University Hospital
Locations (1):
- Ferrara University Hospital, Ferrara, Italy, Italy

REFERENCES:
- [Derived] Straudi S, Severini G, Sabbagh Charabati A, Pavarelli C, Gamberini G, Scotti A, Basaglia N. The effects of video game therapy on balance and attention in chronic ambulatory traumatic brain injury: an exploratory study. BMC Neurol. 2017 May 10;17(1):86. doi: 10.1186/s12883-017-0871-9. PMID 28490322